CLINICAL TRIAL: NCT01802931
Title: An Open Label Study in Healthy Volunteers to Investigate the Effect of Ketoconazole on the Pharmacokinetics of GSK239512
Brief Title: GSK239512 DDI Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 117016
Record Dates: First submitted 2013-01-04; First posted 2013-03-04 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Multiple Sclerosis
Keywords: GSK239512; H3 receptor antagonist; drug-drug interaction; pharmacokinetics; ketoconazole
MeSH Terms: conditions — Multiple Sclerosis | interventions — GSK239512; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Session 1 or Session 2 (Active Comparator): Single dose sessions without ketoconazole co-administration
  Interventions: Drug: GSK239512
- Co-dose Session (Active Comparator): Single dose session with ketoconazole co-administration
  Interventions: Drug: GSK239512; Drug: ketoconazole

INTERVENTIONS:
Drug: GSK239512 — H3 receptor antagonist, potential victim of drug-drug interaction
Drug: ketoconazole — CYP3A4 inhibitor, potential perpetrator of drug-drug interaction
  Arms: Co-dose Session

SUMMARY:
The study will determine the effect of 400 mg once daily of ketoconazole at steady state on the pharmacokinetics of a single oral dose of GSK239512 in young healthy volunteers. Ketoconazole is a strong inhibitor of CYP3A4, which is involved in metabolism of drugs. A two-cohort design will be applied with cohort 1 aimed at providing a first estimate of the interaction potential of GSK239512 and ketoconazole in terms of pharmacokinetic parameters in a small number of subjects. Data from Cohort 1 will inform the decision of which dose to use in Cohort 2, in which a larger number of subjects will be exposed to GSK239512 without and with ketoconazole. The target maximum exposure is aimed to be similar to the exposure by a single dose of 80 mcg of GSK239512 without CYP3A4 inhibition. In summary, the results from this study will help to estimate the maximum increase in exposure of GSK239512 during concomitant use of strong CYP3A4 inhibitors and will help define the subsequent dosing strategy around GSK239512 and co-medications with potential to inhibit CYP3A4.

ELIGIBILITY:
Inclusion Criteria:

1. Male between 18 and 45 years of age inclusive, at the time of signing the informed consent.
2. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
3. ALT, alkaline phosphatase and bilirubin < or = 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
4. QTcF < 450 msec.
5. Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until 1 month post-last dose of GSK239512.
6. Body weight > 50 kg, and body mass index (BMI) between 19.0 - 29.9 kg/m2 inclusive.
7. Capable of giving informed consent and can comply with the study requirements and timetable.

Exclusion Criteria:

1. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
2. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
3. A positive pre-study drug/alcohol screen.
4. A positive test for Human Immunodeficiency Virus (HIV) antibody.
5. History of alcohol consumption exceeding, on average, 21 drinks/week for men (1 drink = 100 mL of wine or 240 mL of beer or 30 mL of hard liquor in Australia) within 6 months of the first dose of study medication.
6. History of smoking cigarettes or using tobacco products or any nicotine-containing products (including nicotine patches) within 3 months of screening.
7. The subject has participated in a clinical trial and has received an investigational product within 30 days or 5 half lives (whichever is longer) prior to the first dosing day in the current study.
8. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
9. Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
10. History of sensitivity to ketoconazole, or to the excipients contained in GSK239512 or Nizoral, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
11. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
12. Unwillingness or inability to follow the procedures outlined in the protocol.
13. Subject is mentally or legally incapacitated.
14. Have used the following medications within the last 30 days or 5 half-lives (whichever is longer) prior to screening and are not able to discontinue use throughout participation in the clinical trial:

    * Any CNS stimulants (e.g., modafinil, dexamphetamine, methylphenidate).
    * Known potent P-glycoprotein inhibitors (e.g. itraconazole, ketoconazole, cyclosporin, loperamide, diltiazem, verapamil, spironolactone, quinidine, bepridil, quinine, carvedilol).
    * Known potent inhibitors or inducers of the CYP3A4 enzyme (see Appendix 3).
    * CNS-penetrant antihistamines (e.g. bromopheniramine, chlorpheniramine, clemastine, diphenhydramine, hyrdoxyzine)
    * Any other medicines that are contraindications of Nizoral (see Appendix 4).
15. Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
16. The subject has a history of significant psychiatric illness.
17. Presence or history of hallucinations that, in the judgement of the investigator, may increase the safety risk to the subject.
18. At risk of suicide, as indicated by:

    * A documented history of attempted suicide or significant suicidal ideation during the 6 months preceding the screening visit, OR
    * If in the investigator's judgment the subject is at risk of a suicide attempt based on the screen visit assessment, including the C-SSRS.
19. Diagnosis of any type epilepsy
20. Night shift workers within 4 weeks of first dosing
21. Presence of significant and routine sleep disturbance that has a negative impact on quality of life that, in the judgement of the investigator, may increase the risk of tolerability issues during dose escalation.

    * Examples of significant sleep disturbances may be: severe insomnia, nocturnal wandering, confusion, disorientation, agitation, or vivid dreams.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2013-01-07 (Actual); Primary Completion 2013-04-15 (Actual); Study Completion 2013-04-15 (Actual)

PRIMARY OUTCOMES:
AUC of GSK239512 | Predose and up to 120 hour post dose of GSK239512
Cmax of GSK239512 | Predose and up to 120 hour post dose of GSK239512

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 117016 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/117016?search=study&search_terms=117016#rs
- Available data/document: Dataset Specification: 117016 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 117016 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 117016 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 117016 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 117016 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 117016 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 117016 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register